CLINICAL TRIAL: NCT07253402
Title: MIcrobiota-Guided RAdiotherapy for Head and Neck Cancer. (MIGRHAN)
Brief Title: Microbiota-guided Radiotherapy for Head and Neck Cancer
Acronym: MIGRAHN
Status: Recruiting | Type: Observational
Sponsor: Fondazione IRCCS Istituto Nazionale dei Tumori, Milano (Other)
Responsible Party: Sponsor
Other Study IDs: INT 84/25
Record Dates: First submitted 2025-11-19; First posted 2025-11-28 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-10

CONDITIONS: Head and Neck Cancer
Keywords: Oral microbiota; Radiotherapy; Tumour control; Oral mucositis; Head and Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms; Stomatitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Saliva samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Radiation: External beam radiotherapy for head and neck cancer — Patients will receive radiotherapy for head and neck cancer and possible concomitant chemotherapies as foreseen by international guidelines. No modification of standard regimens is considered. Intensity-modulated radiotherapy (IMRT) treatment will be administered using X-ray photons with energies ≥6 MV, with daily setup verification performed through IGRT techniques in accordance with institutional standards. Radiotherapy will be delivered with either conventional fractionation or a moderately accelerated hypofractionated schedule (≤2.2 Gy per fraction), with total prescribed doses of up to 70 Gy (2 Gy-equivalent) in the definitive setting, or 54-66 Gy (2 Gy-equivalent) in the postoperative setting. The selection of irradiation targets and dose constraints for organs at risk (OARs) will follow institutional guidelines. OARs will be delineated in accordance with recent international recommendations [Brouwer CL, Radiotherapy and Oncology, 2015].

SUMMARY:
Head and neck cancer (HNC) is the sixth most common cancer worldwide. Therapeutic outcomes for HNC remain unsatisfactory and heterogeneous, with 5-year survival rates ranging from 28% to 67% overall. Moreover, HNC patients experience side effects during treatment, including inflammation and ulceration of the oral mucosa caused by radiation or cytotoxic agents (oral mucositis), which represents a limiting factor for both the escalation of radiotherapy dosage and the duration of treatment.

Several observational studies have highlighted statistical associations between the oral microbiota and numerous factors related to HNC and its therapeutic course. The working hypothesis of this study is that it is possible to establish causal relationships between the functional traits of the human oral microbiota and the effectiveness of radiotherapy in HNC treatment, directly from the analysis of data collected in observational cohorts, by leveraging the statistical framework of causal inference.

The oral microbiota of HNC patients enrolled in the study will be characterised through metagenomic sequencing of saliva samples collected from each patient, at radiotherapy-baseline, at 2 weeks from radiotherapy start and at radiotherapy end.

Main Objectives of the Study:

* Creation of a dataset of the oral microbiota in HNC patients, including both bacterial and viral components, as well as data linked to treatment effectiveness and side effects.
* Estimation of the causal effect of the functional traits of the oral microbiota on the modulation of radiotherapy in HNC.
* Development of predictive models for local tumour control and for oral mucositis, based on the oral microbiota of HNC patients.

Clinical Relevance:

The causal relationships inferred between the functional/metabolic traits of the microbiota and radiotherapy effectiveness will help build interpretable predictive models and reveal strategies to reprogram the microbiota functionality of patients with head and neck cancer. This will increase the likelihood of tumour eradication or control while reducing the risk of radiation-induced side effects.

DETAILED DESCRIPTION:
The research question addressed by this study is the need to bridge the current gap in understanding the role of the microbiota, as well as potential microbiota-targeted therapies such as antibiotic use, in the treatment of head and neck cancer (HNC). The working hypothesis is that causal relationships can be established between the functional traits of the human oral microbiota and the effectiveness of radiotherapy for HNC, using the statistical framework of causal inference. Identifying this causal knowledge is essential to design and implement microbiota-guided radiotherapy, where the patient's oral microbiota is profiled prior to treatment and evaluated against the risk of developing oral mucositis and/or experiencing unfavorable outcomes. From a microbiota-based perspective, assessing whether different radiotherapy plans may result in tolerable or intolerable side effects would be crucial for developing personalized radiotherapy programs that could enhance tumor control. Furthermore, since this study involves functional metagenomic analysis of the microbiota, it will be possible to infer the mechanisms through which the microbiota modulates radiotherapy and to exploit these insights for the design of new microbiota-based clinical strategies. Such strategies may include administration of specific nutritional supplements, antibiotics, or probiotics to optimise therapy tolerance and improve treatment outcomes.

Study design and setting: MIGRHAN is a single-institution, prospective observational cohort study with an expected total duration of approximately six years. At least 96 consecutive patients with head and neck cancer referred for curative radiotherapy will be enrolled over a 36-month period. Their treatment, toxicity monitoring, and follow-up (3 years) will follow routine clinical practice in accordance with national and international guidelines. Recruitment will take place exclusively at Fondazione IRCCS Istituto Nazionale dei Tumori, Milan, with patient enrollment starting in September 2025 and planned completion by October 2031.

Study workflow: Before enrollment, patients will provide written informed consent. Baseline assessments (from -28 days to treatment start) will include demographic data, medical history, dental evaluation, clinical examination, laboratory tests (blood tests, urinalysis, thyroid function, coagulation), radiological imaging (CT scan, multiparametric MRI, whole body FDG-PET/CT or bone scan), and collection of a saliva sample for microbiota profiling. During radiotherapy, weekly clinical evaluations, toxicity assessments following CTCAE v5.0, and patient questionnaires will be conducted, alongside repeated laboratory analyses and collection of dosimetric treatment data (DICOM-RT). At the end of radiotherapy and during follow-up visits (3, 6, and 12 months), patients will undergo repeat clinical evaluations, imaging (MRI, CT, PET/CT or bone scan as indicated), laboratory tests, and additional saliva collections. Long-term follow-up will include survival assessment up to three years post-treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* ECOG Performance Status ≤ 3.
* Histological diagnosis of squamous cell carcinoma, undifferentiated carcinoma, epithelial glandular and non-glandular carcinoma (including adenoid cystic carcinoma, adenocarcinoma, mucoepidermoid carcinoma, neuroendocrine carcinoma, etc.) originating from the oral cavity, oropharynx, nasopharynx, hypopharynx, larynx, salivary glands, paranasal sinuses, or from an unknown primary site.
* Stage III-IV non-metastatic disease for pharyngeal, laryngeal, or unknown-primary tumors, according to AJCC 7th edition. Patients with stage III-IV tumors of salivary gland or paranasal sinus origin, and patients with stage I-II pharyngeal or laryngeal tumors, will only be included if prophylactic irradiation of cervical lymph node stations is indicated and/or if the oral and oropharyngeal mucosa as well as swallowing-related structures are included within the irradiated volume.
* Indication for treatment in either definitive or adjuvant settings, with or without systemic therapy (concurrent systemic therapy, with or without prior neoadjuvant chemotherapy, permitted. Adjuvant systemic therapy is allowed for selected advanced stages of pharyngeal carcinoma, according to institutional guidelines).
* Formal acceptance of study participation requirements (written informed consent).

Exclusion Criteria:

* Prior radiotherapy to the head-neck region.
* Presence of connective tissue disorders (e.g., lupus erythematosus or scleroderma) or synchronous head and neck malignancies, except for superficial skin cancers or surgically treated carcinoma in situ not requiring radiotherapy or systemic therapy.
* Absence of formal acceptance of study participation requirements (written informed consent).
* Indication for treatment exclusively in the postoperative setting.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing external beam radiotherapy for head and neck cancer at Fondazione IRCCS Istituto Nazionale dei Tumori di Milano.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-10-15 (Actual); Primary Completion 2031-10-30 (Estimated); Study Completion 2031-10-30 (Estimated)

PRIMARY OUTCOMES:
Locoregional tumour control | 1 year following radiotherapy end
  The primary endpoint is local tumor control at 12 months of follow-up, considering both partial and complete responses as defined by the oncological RECIST 1.1 radiological criteria. Tumor volume analysis from MRI imaging between pre-RT and 3 months post-RT will be used to quantify tumor volume reduction (shrinkage) in patients undergoing curative radiotherapy alone. Tumor volume analysis from MRI imaging at 3, 6, and 12 months post-RT will be used to quantify tumor volume recurrence.

SECONDARY OUTCOMES:
Acute toxicity | <8 weeks from radiotherapy end
  Toxicity assessment will be performed by the radiation oncologist in accordance with CTCAE v.5.0 recommendations, through the completion of questionnaires and clinical evaluation. Clinician-reported outcomes (CROs), collected weekly during radiotherapy, will be used to define longitudinal descriptors of the onset and severity of treatment-related side effects. Descriptors of interest will include mean mucositis grade, incidence of grade ≥3 mucositis, and maximum mucositis grade. In addition to CRO-based descriptors, the feasibility of defining quantitative toxicity descriptors will be explored through the analysis of normal tissues on MRI images by extracting textural features.

OTHER OUTCOMES:
Progression-free survival (PFS) | 3 years from radiotherapy end
  Progression-free survival (PFS) will be defined as the time interval from the start of treatment to the occurrence of either the first documented disease progression or death from any cause, whichever occurs first.

CONTACTS AND LOCATIONS:
Overall Officials: Jacopo Iacovacci, PhD, Principal Investigator — Fondazione IRCCS Istituto Nazionale dei Tumori di Milano; Nicola A Iacovelli, MD, Study Director — Fondazione IRCCS Istituto Nazionale dei Tumori di Milano; Loris DeCecco, PhD, Study Director — Fondazione IRCCS Istituto Nazionale dei Tumori di Milano
Locations (1):
- Fondazione IRCCS Istituto Nazionale dei Tumori di Milano, Milan, Milan, Italy

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-09-05): https://cdn.clinicaltrials.gov/large-docs/02/NCT07253402/Prot_SAP_000.pdf